CLINICAL TRIAL: NCT03711617
Title: The Association Between Uremic Toxins and Outcomes and Comorbidities in Patients With CKD
Brief Title: Uremic Toxins and Outcomes in Chronic Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Ding Feng, Director of Devision of Nephrology, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: CKD-toxins
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; uremic toxin; prognosis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine,serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CKD-ND: patients with non-dialysis CKD
- CKD-MHD: patients with maintenance hemodialysis

SUMMARY:
The aim of this cohort study is:

To investigate the etiology and epidemiology of comorbidities in CKD; To find out risk factors associated with the mortality of CKD; To find out uremic toxins which are related to the mortality and comorbidities of CKD; To focuse on the association between uremic toxins and inflammation, oxidative stress and nutritional status in CKD.

DETAILED DESCRIPTION:
To investigate the etiology and epidemiology of comorbidities in CKD; To find out risk factors associated with the mortality of CKD; To find out uremic toxins which are related to the mortality and comorbidities of CKD; To focuse on the association between uremic toxins and inflammation, oxidative stress and nutritional status in CKD.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old;
* clinically diagnosed with chronic kidney disease, according K/DOQI criteria.

Exclusion Criteria:

* acute kidney injury
* history of kidney injury <3 months
* malignancy
* pregnancy
* incomplete clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CKD patients from hospitals
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 5 years

SECONDARY OUTCOMES:
comorbidities | 5 years
  CVD,mortality,hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ding, PhD, Study Chair — Division of Nephrology, Shanghai Ninth People's Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China